CLINICAL TRIAL: NCT07153679
Title: Efficacy and Safety of a 1064-nm Nd:YAG Picosecond Laser Versus a 1927-nm Fractional Thulium Laser for Atrophic Acne Scars in Asian Skin: A Randomized, Split-Face, Evaluator-Blinded Trial.
Brief Title: Efficacy and Safety of a 1064-nm Nd:YAG Picosecond Laser Versus a 1927-nm Fractional Laser for Atrophic Acne Scars.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Weihui Zeng, professor, Second Affiliated Hospital of Xi'an Jiaotong University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 2021013
Record Dates: First submitted 2025-08-26; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Acne Scar; Acne Scars - Atrophic

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1064-nm Nd:YAG Picosecond Laser Group (Experimental): 1064-nm Nd:YAG Picosecond Laser Device (Picocare 450, WONTECH, Daejeon, South Korea)
  Interventions: Device: 1064-nm Nd:YAG Picosecond Laser
- 1927-nm Fractional Thulium Laser Group (Experimental): 1927-nm Fractional Thulium Laser Device (Lavieen, WONTECH, Daejeon, South Korea)
  Interventions: Device: 1927-nm Fractional Thulium Laser

INTERVENTIONS:
Device: 1064-nm Nd:YAG Picosecond Laser — Treatment was performed using 1064 nm Nd:YAG microlens array picosecond laser (Picocare 450, WONTECH, Daejeon, South Korea). Received three treatments, with a 4-week interval between each treatment.
  Arms: 1064-nm Nd:YAG Picosecond Laser Group
Device: 1927-nm Fractional Thulium Laser — Treatment was performed using 1927-nm thulium fractional laser (Lavieen, WONTECH, Daejeon, South Korea). Received three treatments, with a 4-week interval between each treatment.
  Arms: 1927-nm Fractional Thulium Laser Group

SUMMARY:
Atrophic acne scars are common disfiguring skin problems, especially in the Asian population prone to Post-inflammatory Hyperpigmentation (PIH), and their treatment is highly challenging. 1064 nm microlens array picosecond laser (P-MLA) based on optomechanical effect and 1927 nm segmented thulium laser (FTL) based on photothermal effect are two emerging therapeutic techniques, but there is a lack of strict clinical evidence for direct comparison in the Asian population. This study aims to directly compare the clinical efficacy, safety and tolerability of 1064 nm P-MLA and 1927 nm FTL in the treatment of atrophic acne scars in the Asian population through a randomized, half-face controlled, evaluator blind trial.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 40.
* Symmetrical atrophic acne scars on both sides of the face.

Exclusion Criteria:

* Uncontrolled active acne.
* Pregnant and lactating women.
* Infectious skin diseases at the treatment site.
* Have taken retinoid drugs orally within the past 6 months.
* Photosensitive individuals or those who have used photosensitive drugs within 2 weeks.
* Keloid constitution.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
ECCA grading scale | Baseline and 20 weeks.
  Scar shape: U-shaped sharp-edged scars (2-4 mm) = 20 points, irregular U-shaped (>4 mm) = 25 points. Scar number: 0 scars = 0, ≤5 scars = 1, 6-20 scars = 2, >20 scars = 3. ECCA score = Shape score × Number score. Higher score = more severe scarring.
GAIS score | Baseline and 20 weeks.
  GAIS score: 1 = 0%-25% improvement; 2 = 26%-50%; 3 = 51%-75%; 4 = 76%-100%. Higher score = better improvement.

SECONDARY OUTCOMES:
Melanin Index | Baseline and 20weeks.
  Utilizing the DermaLab® Combo (Cortex Technology)
Erythema Index | Baseline and 20 weeks.
  Utilizing the DermaLab® Combo (Cortex Technology)
Transepidermal Water Loss | Baseline and 20 weeks.
  Utilizing the DermaLab® Combo (Cortex Technology)

CONTACTS AND LOCATIONS:
Locations (1):
- The second affiliated hospital of Xi'an Jiaotong University, Xi’an, Shanxi, China

IPD SHARING:
Plan to Share IPD: No